CLINICAL TRIAL: NCT06052345
Title: Chemotherapy(paclitaxel)-induced Polyneuropathy in Breast Cancer As Part of the REBECCA Project (REsearch on BrEast Cancer Induced Chronic Conditions Supported by Causal Analysis of Multi-source Data)
Brief Title: Paclitaxel-induced Polyneuropathy in Breast Cancer: Early Detection, Risk Factors, Quality of Life and Lifestyle Outcomes
Acronym: CIPN-REBECCA
Status: Recruiting | Type: Observational
Sponsor: Theodoros Foukakis (Other)
Collaborators: Karolinska Institutet (Other); Centre for Research and Technology Hellas (CERTH) (Unknown)
Responsible Party: Sponsor-Investigator, Theodoros Foukakis, Senior Consultant, Associate Professor of Oncology, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Other Study IDs: 2022-04453-01; 965231 (Other Grant/Funding Number: European Union's Horizon 2020 research and innovation programme)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms; Breast Cancer; Early-stage Breast Cancer; Non-Metastatic Breast Carcinoma; Polyneuropathy Due to Drugs; Polyneuropathy; Drug; Chemotherapy-induced Peripheral Neuropathy; Quality of Life
Keywords: Paclitaxel-induced polyneuropathy; Antineoplastic Agents; Plant Alkaloids; Paclitaxel; Adjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Polyneuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and skin samples will be taken in different timepoints of the study as described in the protocol. Specifically, from each patient at least 10 ml of blood will be collected and 2 skin samples (3 mm wide, 2-3 mm deep)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CIPN group: Breast cancer patients that developed strong CIPN symptomatology at post-treatment evaluation (4 weeks after the end of therapy)
  Interventions: Device: Garmin smartwatch; Other: REBECCA Mobile application; Other: REBECCA PC plug-in
- No-CIPN group: Breast cancer patients that developed mild-to-no CIPN symptomatology at post-treatment evaluation (4 weeks after the end of therapy)
  Interventions: Device: Garmin smartwatch; Other: REBECCA Mobile application; Other: REBECCA PC plug-in

INTERVENTIONS:
Device: Garmin smartwatch — * Physical activity (Activity sessions, type and length of activity, activity intensity estimations)
  * Meal detection and meal characteristics (accelerometry and gyroscope data)
  * Oxygen saturation (pulse oximetry)
  * Number of steps (pedometer)
  * Stress level indicators (based on heart-rate analytics)
  * Sleep patterns (sleep and wake-up time, sleep quality)
Other: REBECCA Mobile application — * GPS positioning (daily location change patterns through pathway analysis and Point-of-interest analysis based on type-of-location automatic detection)
  * Self-reports from patients and companions reports on mental and physical health, as well as periodic quality of life evaluations3
  * Patient self-uploaded pictures of meals (for evaluation of nutritional habits) and living environment stressors (for evaluation of living environment and self-perceived stressor analysis)
Other: REBECCA PC plug-in — * the developed plug-in monitors online activity, collecting anonymized data from web-browsers (Chrome) and social media (Facebook, Youtube and Instagram).
  * These are relevant to current and historical data on: i) keywords in searches, ii) types of websites visited, iii) reactions to posts, iv) participation in online groups, v) types of bookmarked websites

SUMMARY:
This is a single center prospective observational cohort study that aims to:

* examine and identify possible risk and susceptibility factors for the incidence and progression of chemotherapy-induced polyneuropathy (CIPN) in female patients primarily operated for early non-metastatic breast cancer who will receive adjuvant chemotherapy containing paclitaxel
* test different neurophysiological methods for early detection of CIPN
* explore changes that underlie the development of CIPN in relation to clinical presentations, neurophysiological assessment, including measures of small nerve fiber dysfunction, and possible biochemical, metabolic and genetic associations
* explore the effects of CIPN in the patient's lifestyle and quality of life for up to 12 months after the initiation of treatment

DETAILED DESCRIPTION:
The patients who follow the inclusion criteria of the study will be asked to complete:

* a baseline evaluation prior to receiving treatment. This will include a bedside clinical-neurological evaluation, nerve conduction studies (NCS) and quantitative sensory tests of thermal threshold (QST), blood sampling, an oral glucose tolerance test, a skin biopsy, and answering of questionnaires for assessment of symptoms of peripheral neuropathy as well as self-reports on their pre-treatment health and lifestyle status and cancer specific symptomatology
* an on-treatment evaluation 4 weeks after the start of the treatment which will include NCS and QST
* a post-treatment evaluation 4 weeks after the end of treatment which will include the evaluations stated above. During this visit the participants will be provided with the REBECCA lifestyle monitoring system which will include a smartwatch, installation of a mobile app and a PC plugin. The patients will be also asked to fill in some self-rated evaluations as in the pre-treatment period. Researchers, based on the outcomes of the participants, will divide them in two study groups A. CIPN-group and B. No CIPN which will be monitored with the REBECCA monitoring system.
* a final evaluation. This will be performed 8 months after the post-treatment evaluation and it will include clinical-neurological evaluation, nerve conduction studies (NCS) and thermal threshold testing (QST). Additionally, the participants will be requested to fill in the same self-rated evaluations as in the baseline and the post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age of ≥ 18 years
* Newly operated primary breast cancer without metastatic disease receiving adjuvant chemotherapy containing paclitaxel
* No prior chemotherapy other than cyclophosphamide and epirubicin
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Written informed consent
* Able to communicate with investigators, participate in testing and comply with the requirements of the study-protocol

Exclusion Criteria:

* Have received drugs suspected/known to cause peripheral neuropathy
* Have history of acquired or inherited neuropathy or other genetic disease with increased tendency to develop neuropathy
* Have known disturbed glucose metabolism, either diabetes mellitus or impaired glucose tolerance
* Have moderate to severe kidney, liver, lung or heart disease
* Have known symptomatic or other advanced spinal stenosis
* Have known autoimmune disease that potentially cause or contribute to neuropathy
* Have known HIV or active HBV or HCV infections
* Have known paraneoplastic syndrome
* Have known alcohol abuse
* Have known pregnancy or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified as potential candidates and consecutively recruited from the oncology clinic at Karolinska University Hospital in Solna. Eligible candidates are patients who have been primarily operated for early non-metastatic breast cancer and are recommended by the multidisciplinary conference to receive adjuvant chemotherapy containing paclitaxel.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of significant deterioration in neurophysiological parameters including alterations in morphology of small fibers or reduced IENFD (Intraepidermal Nerve Fiber Density) on first follow up visit and development of CIPN | 1 year
  by performing detailed clinical neurophysiological examination and skin biopsies (where IENFD will be quantified) in different timepoints as described in the study protocol
Correlation of abnormal laboratory tests in baseline assessment with development/severity of CIPN | 1 year
Correlation of parameters of NCS, temperature thresholds, and IENFD at baseline screening with development and severity of CIPN | 1 year
Biochemical and metabolic abnormalities prior to paclitaxel treatment and their association with the development of CIPN | 1 year
  by performing blood tests, genotyping and skin biopsies

SECONDARY OUTCOMES:
Calculate and compare the false negative and false positive rate of CIPN in every used method during follow up | 1 year
Association of altered scoring in different questionnaires (Fact/GOG-Ntx, SFN-SIQ) and different examinations (UENS) with the presence and severity of CIPN | 1 year
Evaluation of whether specific genotypes of breast cancer and higher or lower levels of different proteins are related with higher incidence rate and severity of CIPN | 2 years
  by extracting DNA from blood samples and performing subsequent genotyping using SNP-array and GWAS. Also, by using proteomics analysis in blood samples and measure plasma levels of different proteins.
Study any correspondence between deterioration of QoL indicated by REBECCA monitoring system and standardized patient self-reported measures with diagnosed CIPN after implementation of different methods during follow up | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Foukakis, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Solna, Stockholm County, Sweden

REFERENCES:
- See also: REBECCA stands for REsearch on BrEast Cancer induced chronic conditions supported by Causal Analysis of multi-source data and aims to tap into the potential of Real-World Data to support clinical research and to improve existing clinical work — https://rebeccaproject.eu/